CLINICAL TRIAL: NCT06018428
Title: A Phase 2a, Randomized, Double-blind, Placebo-Controlled, Proof-of-Concept Trial With Part B and Open-label Extension of Bempikibart (ADX-914) for the Treatment of Severe Alopecia Areata (SIGNAL-AA)
Brief Title: A Phase 2a Proof-of-Concept Trial of Bempikibart (ADX-914) for the Treatment of Severe Alopecia Areata (SIGNAL-AA)
Acronym: SIGNAL-AA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Q32 Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADX-914-203; SIGNAL-AA (Other: Q32 Bio)
Record Dates: First submitted 2023-08-15; First posted 2023-08-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Alopecia Areata
Keywords: Areata, Alopecia; Alopecia; Dermatitis; Hair Loss; Trichoscopy; Atopic
MeSH Terms: conditions — Alopecia Areata; Alopecia; Dermatitis

STUDY DESIGN:
Masking Description: Part A was double blind-randomized. Part B and OLE are open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: bempikibart (ADX-914) (Experimental): 200mg dose of bempikibart (ADX-914) administered via injection under the skin
  Interventions: Drug: bempikibart (ADX-914)

INTERVENTIONS:
Drug: bempikibart (ADX-914) — Subcutaneous administration of bempikibart (ADX-914)

SUMMARY:
Part A is a randomized, double-blind, placebo-controlled, multi-center Proof-of-Concept (POC) Trial in subjects with severe Alopecia Areata. All participants in Part A have completed participation.

Part B is a multicenter, open-label study to assess the efficacy, safety, and tolerability of bempikibart (ADX-914) in participants with severe Alopecia Areata.

DETAILED DESCRIPTION:
Part A is a Phase IIa, Randomized, Double-blind, Placebo-controlled, multi-center Proof-of-Concept (POC) study in adult subjects with severe Alopecia Areata (AA). Bempikibart (ADX-914) or matching placebo is administered subcutaneously in the clinic setting every 2 weeks for 24 weeks, with follow-up for 12 weeks. Subjects will be randomized 3:1 to drug vs placebo. All participants in Part A have completed participation.

Part B is a multicenter, open-label study comprised of a screening period of up to 4 weeks, a treatment period of 36 weeks, and a follow-up period of 16 weeks, for a total study duration of up to 56 weeks.

Open Label Extension Cohort is a multicenter, open-label extension to assess the long-term efficacy, safety, and tolerability of bempikibart (ADX-914) in participants with severe AA who experienced hair regrowth as participants in Part A of the study. Participants enrolled in the Open Label Extension Cohort will receive bempikibart (ADX-914) for a duration of 6 months followed by a 16-week follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult men and women, aged 18 to 75 years, inclusive, at the time of informed consent.
2. Clinical diagnosis of severe to very severe alopecia areata, defined as the presence of ≥50% total scalp hair loss at screening and baseline as measured by the SALT score.

Key Exclusion Criteria:

1. History of or diagnosis at screening of any another form of alopecia based on assessment by investigator.
2. History (lifetime) or presence of hair transplants.
3. History (lifetime) or presence of micropigmentation of the scalp (Note: Microblading of the eyebrows is permitted).
4. Use of systemic, topical, or device-based therapy for AA.
5. History of, recent, or current clinically serious viral, bacterial, fungal, or parasitic infection or mycobacterial infection or at risk of serious infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Part A: Mean relative percent change in SALT score | 24 Weeks
  Part A: Mean relative percent change in SALT score at 24 weeks compared with baseline
Part B: Mean percent change from baseline in SALT score | 36 weeks
  Part B: Mean percent change from baseline in SALT score at Week 36

SECONDARY OUTCOMES:
Part A: Mean relative percentage change SALT score compared with baseline at Weeks 6,12, and 18. | 18 Weeks
Part A: Mean relative percentage change in SALT score at 24 weeks compared with treatment nadir. | 24 Weeks
Part A: Absolute change in SALT score compared with baseline at Weeks 6, 12, 18, and 24. | 24 Weeks
Part A: Proportion of participants who achieve ≥30% and ≥50% relative reduction in SALT score compared with baseline at Weeks 12, 18, and 24. | 24 Weeks
Part A: Proportion of participants with absolute SALT score ≤5, ≤10, ≤20, and ≤30 at Weeks 12, 18, and 24. | 24 Weeks
Part A: Overall Safety as evaluated by number of adverse events (AEs). | 36 Weeks
Part B: Proportion of participants who achieve ≥50% relative reduction in SALT score compared with baseline at 36 weeks | 36 Weeks
Part B: Mean percent change from baseline in SALT score at Week 52 | 52 Weeks
Part B: Proportion of participants with absolute SALT score ≤20 and ≤30 at Week 36. | 36 Weeks

CONTACTS AND LOCATIONS:
Locations (32):
- United States (27):
  - Scottsdale, Arizona, Scottsdale, Arizona
  - Fayetteville, Arkansas, Fayetteville, Arkansas
  - Hot Springs, Arkansas, Hot Springs, Arkansas
  - Encinitas, California, Encinitas, California
  - Fountain Valley, California, Fountain Valley, California
  - Lomita, California, Lomita, California
  - New Haven, Connecticut, New Haven, Connecticut
  - Miami, Florida, Miami, Florida
  - Tampa, Florida, Tampa, Florida
  - Clarksville, Indiana, Clarksville, Indiana
  - Bowling Green, Kentucky, Bowling Green, Kentucky
  - Burlington, Massachusetts, Burlington, Massachusetts
  - Troy, Michigan, Troy, Michigan
  - Warren, Michigan, Warren, Michigan
  - New York, New York, New York, New York
  - Wilmington, North Carolina, Wilmington, North Carolina
  - Bexley, Ohio, Bexley, Ohio
  - Clinical Trials, Canton, Ohio
  - Mason, Ohio, Mason, Ohio
  - Mayfield Heights, Ohio, Mayfield Heights, Ohio
  - Portland, Oregon, Portland, Oregon
  - Austin, Texas, Austin, Texas
  - Frisco, Texas, Frisco, Texas
  - Houston, Texas, Houston, Texas
  - San Antonio, Texas, San Antonio, Texas
  - Jordan, Utah, Jordan, Utah
  - Spokane, Washington, Spokane, Washington
- Canada (5):
  - Clinical Trials, Calgary, Alberta
  - Clinical Trials, Winnipeg, Manitoba
  - Clinical Trials, Oakville, Ontario
  - Clinical Trials, Peterborough, Ontario
  - Clinical Trials, Waterloo, Ontario